CLINICAL TRIAL: NCT06293430
Title: Registry on Luma Vision's VERAFEYE System in Catheter Ablation and Left Atrial Appendage Closure Procedures
Brief Title: Registry on Luma Vision's VERAFEYE System (ENLIgHT)
Acronym: ENLIgHT
Status: Not yet recruiting | Type: Observational
Sponsor: LUMA Vision Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ENLIgHT-P002
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Atrial Fibrillation; Left Atrial Appendage Closure; Atrial Arrhythmia
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: VERAFEYE System — VERAFEYE system guidance will be used on all patients undergoing AF ablation and/or LAAC procedures.

SUMMARY:
The objective of the study is to compile real-world data on the use of the VERAFEYE System in standard of care atrial fibrillation (AF) ablation procedures and left atrial appendage closure (LAAC) procedures.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject is 18 years of age or of legal age to give informed consent specific to state and national law at the time of consent
* Subjects is indicated for an atrial fibrillation ablation and/or a left atrial appendage closure procedure with the VERAFEYE System as navigation and imaging system, per physician discretion;
* Subject is able to understand and willing to provide written informed consent
* Subject is able and willing to complete all study assessments at an approved clinical investigational center

Key Exclusion Criteria:

* Subjects who have undergone a previous cardiac ablation for the treatment of PAF/LAA Closure
* Subject where placement of VERAFEYE Imaging Catheter is technically not feasible per physician discretion
* Pregnant women or women who plan to become pregnant during the course of their participation in the study (women should either be of non- childbearing potential at the time of enrolment (as documented in the medical file) or have a negative pregnancy test within the previous 7 days prior to the procedure)
* Unrecovered/unresolved Adverse Events from any previous invasive procedure
* Subjects who are currently enrolled in another study (except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the investigator's general patient population. Subjects considered for participation in this study will be entitled to undergo a standard of care PAF ablation and/or LAAC procedure with the VERAFEYE System.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-10-15 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Acute procedural success rates during the index procedure | During the procedure
  A procedure will be defined as successful if all the following conditions occur during the case:
  * ability to create a 3D anatomical model with the VERAFEYE System and
  * completion of the necessary ablation applications for PAF/LAA Closure using the 3D anatomical model created with the VERAFEYE System

IPD SHARING:
Plan to Share IPD: No